CLINICAL TRIAL: NCT01761435
Title: Randomized, Comparative and Prospective Clinical Trial Evaluating Efficacy and Safety of a Dose of Seasonal Flu Vaccine Compared to Two Doses of Vaccine for Prevention of Influenza in Solid Organ Transplant Recipients
Brief Title: Clinical Trial Evaluating Efficacy and Safety of One Dose Versus Two Doses of Influenza Vaccination
Acronym: TraNsgripe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Collaborators: Spanish Network for Research in Infectious Diseases (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TraNsgripe1-2
Record Dates: First submitted 2012-12-13; First posted 2013-01-04 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Infection in Solid Organ Transplant Recipients
Keywords: Influenza; Solid Organ Transplant Recipients
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine, second administration after 5 weeks (Experimental): Drug: Influenza vaccine (split virion, inactivated) suspension for injection 0.5ml at the baseline and 5 weeks after the first one.
  Interventions: Biological: Influenza vaccine
- Influenza vaccine (Active Comparator): Drug: Influenza vaccine (split virion, inactivated) suspension for injection 0.5ml at the baseline.
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Patients will be randomized at 1:1 rate and open label fashion, according to centers, and time elapsed since transplant and type of organ transplanted to one of this two interventions :
  A arm (usual treatment): Influenza vaccine (split virion, inactivated) suspension for injection 0.5ml at the baseline.
  B arm (experimental branch): Influenza vaccine (split virion, inactivated) suspension for injection 0.5ml at the baseline and 5 weeks after the first dose.
  The follow-up of both arms will be at 5, 10 and 15 weeks and one year after the baseline.

SUMMARY:
Randomized, multicenter, open label trial to compare safety and efficacy of two doses stationary flu vaccination vs one doses in Solid Organ Transplant Recipients.

DETAILED DESCRIPTION:
The purposes of this study are:

1. Evaluate the efficacy and safety of a double dose of seasonal flu vaccine compared to a single dose.
2. Determine the specific cellular immune response produced after the first and second vaccine doses of seasonal flu vaccine by in vitro stimulation of specific memory cells (A and B flu viruses).
3. Evaluate the humoral immune response produced after one dose vs two doses of seasonal flu vaccine by the measure of serum antibody levels.
4. Evaluate clinical efficacy of stationary flu vaccine in solid organ transplant recipients.
5. Evaluate a long term cellular and humoral response(1 year) of seasonal flu vaccine.
6. Characterize the genetic expression profile of immune response after the flu vaccine in solid organ transplant recipients by means of a genetic sub-study.
7. Characterize the flu vaccine effect (one dose and two doses) through the antibody anti-HLA(human leukocyte antigen), and its influence on the rejection rate in solid organ transplant recipients, by means of immunologic sub-study.

ELIGIBILITY:
Inclusion Criteria:

1. Solid organ transplant recipient.
2. 16 years or older.
3. More than 30 days after transplantation.
4. Negative pregnancy test for women of childbearing potential
5. The patient must give informed consent

Exclusion Criteria:

1. No written informed consent.
2. Acute rejection within 15 days prior to vaccination.
3. Pregnancy.
4. Hypersensitivity to the active substance, any of the excipients and waste, for example: eggs, egg albumin, chicken proteins.
5. History of a previous serious reaction to immunization (eg Guillain-Barré syndrome).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates | At 5, 10, 15 weeks, and 12 months after the first vaccine dose
  Difference in seroconversion rates in both treatment groups at 5, 10, 15 weeks, and 12 months after the first vaccine dose (percent of patients with 4 x increase in the pre-vaccination titers).

SECONDARY OUTCOMES:
Postvaccination antibody titers | At 5, 10, 15 weeks, and 12 months after the first vaccine dose.
  Geometric average postvaccination antibody titers and rate of increase between pre-and post-vaccination geometric mean, post-vaccination seroprotection rate (or percentage of individuals with a titer 1 / 40 as measured by RIH).
Safety. | At 5, 10, 15 weeks, and 12 months after the first vaccine dose
  Occurrence of grade 3 or 4 toxicity, death, hospitalization, retransplantation, acute rejection and chronic rejection
Efficacy | At 5, 10, 15 weeks, and 12 months after the first vaccine dose
  Detection of clinical cases of influenza following immunization. Nasal swabs to confirm infection with influenza virus by RT-PCR (Reverse transcription polymerase chain reaction).
Antibody anti-HLA | At 5, 10, 15 weeks, and 12 months after the first vaccine dose
  Characterize the flu vaccine effect (one dose and two doses) through the antibody anti-HLA levels, ant its influence on the rejection rate in solid organ transplant recipients, by means of immunologic sub-study.
Cellular response | At 5, 10, 15 weeks, and 12 months after the first vaccine dose
  Determination of the T cells specific immune response measured by production of INFg, IL-2 and IL-4 in the cytoplasm of CD4+ and CD8 + (mononuclear cells) specific for influenza virus by direct immunofluorescence and flow cytometry analysis.
Clinical complications | At 5, 10, 15 weeks, and 12 months after the first vaccine dose
  Clinical severity (hospitalization, ICU admission, death, rejection). Time to clinical stability will be register.

CONTACTS AND LOCATIONS:
Overall Officials: Julian De la Torre Cisneros, PhD, Principal Investigator — COMPLEJO HOSPITALARIO REGIONAL REINA SOFÍA; Francisco López Medrano, PhD, Principal Investigator — Hospital Universitario 12 de Octubre; Patricia Muñoz García, PhD, Principal Investigator — HOSPITAL GENERAL GREGORIO MARAÑÓN; Jesús Fortun Abete, PhD, Principal Investigator — Hospital Universitario Ramon y Cajal; Joán Gavaldà Santapau, PhD, Principal Investigator — HOSPITALS VALL D'HEBRON; Jordi Carratalá Fernández, PhD, Principal Investigator — Hospital Universitari de Bellvitge; Asunción Moreno Camacho, PhD, Principal Investigator — Hospital Clinic i provincial de Barcelona; José Miguel Montejo Baranda, PhD, Principal Investigator — HOSPITAL UNIVERSITARIO DE CRUCES; Marino Blanes Julia, PhD, Principal Investigator — Hospital Universitario La Fe; Alejandro Suarez Benjumea, PhD, Principal Investigator — COMPLEJO HOSPITALARIO REGIONAL VIRGEN MACARENA; Carmen Fariñas Álvarez, PhD, Principal Investigator — Hospital Universitario Marqués de Valdecilla; Maria Elisa Cordero Matia, PhD, Principal Investigator — Hospital Universitario Virgen del Rocio
Locations (12):
- Spain (12):
  - Hospital Clinic Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona, Barcelona
  - Hospital Universitario de Cruces, Bilbao, Bilbao
  - Hospital Universitario Masqués de Valdecilla, Santander, Bilbao
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital General Gregorio Marañon, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario 12 Octubre, Madrid, Madrid
  - Hospital Vall d'Hebron, Madrid, Madrid
  - Hospital Universitario Virgen del Rocío, Seville, Sevilla
  - Hospital Regional Virgen de la Macarena, Seville, Sevilla
  - Hospital la Fe de Valencia, Valencia, Valencia

REFERENCES:
- [Derived] Demetz G, Laux M, Scherhag A, Hoekstra T, Suttorp MM, Dekker F, Roest M, Marcus-Kalish M, Mittelman M, Ott I. The influence of Erythropoietin on platelet activation, thrombin generation and FVII/active FVII in patients with AMI. Thromb J. 2014 Aug 28;12:18. doi: 10.1186/1477-9560-12-18. eCollection 2014. PMID 25228850
- [Derived] Martinez-Atienza J, Rosso-Fernandez C, Roca C, Aydillo TA, Gavalda J, Moreno A, Montejo JM, Torre-Cisneros J, Farinas MC, Fortun J, Sabe N, Munoz P, Blanes-Julia M, Suarez-Benjumea A, Lopez-Medrano F, Perez-Romero P, Cordero E; TRANSGRIPE 1-2 Study Group. Efficacy and safety of a booster dose of influenza vaccination in solid organ transplant recipients, TRANSGRIPE 1-2: study protocol for a multicenter, randomized, controlled clinical trial. Trials. 2014 Aug 28;15:338. doi: 10.1186/1745-6215-15-338. PMID 25168918
- See also: The Spanish Network for the Research in Infectious Diseases (REIPI) is based in research groups of high standards and professional level. REIPI´s aim is to generate scientific knowledge in the field of the infectious diseases, in areas ranging from basic — http://www.reipi.org/